CLINICAL TRIAL: NCT02975310
Title: Endoscopic Polypectomy Performed In Clinic for Chronic Rhinosinusitis With Polyps: The EPIC Randomised Controlled Trial
Brief Title: In-clinic Endoscopic Polypectomy for Chronic Sinusitis With Nasal Polyps
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Ottawa Hospital Research Institute (Other)
Collaborators: Canadian Institutes of Health Research (CIHR) (Other Government); Medtronic (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: CTO-0801
Record Dates: First submitted 2016-11-17; First posted 2016-11-29 (Estimated); Last update posted 2025-12-30 (Actual); Status verified 2025-12

CONDITIONS: Sinusitis; Nasal Polyps
MeSH Terms: conditions — Sinusitis; Nasal Polyps | interventions — Ambulatory Care Facilities; Anesthesia, General; Anesthesia

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Endoscopic polypectomy in clinic (EPIC) (Experimental): Patients assigned to this arm of the study will undergo the In Clinic Polypectomy Performed in Clinic
  Interventions: Procedure: Endoscopic polypectomy in clinic (EPIC); Other: Local and topical anesthesia
- Endoscopic Sinus Surgery (ESS) (Active Comparator): Patients assigned to this arm will undergo endoscopic sinus surgery (ESS),
  Interventions: Procedure: Endoscopic Sinus Surgery (ESS); Other: General Anesthesia

INTERVENTIONS:
Procedure: Endoscopic polypectomy in clinic (EPIC) — The experimental intervention is endoscopic polypectomy performed in clinic (EPIC) where nasal polyps are removed using a microdebrider under local and topical anesthesia in the outpatient clinic.
  Arms: Endoscopic polypectomy in clinic (EPIC)
Procedure: Endoscopic Sinus Surgery (ESS) — The control intervention is endoscopic sinus surgery (ESS), a minimally invasive procedure that is the current standard that involves polypectomy with a microdebrider as well as sinus ostia enlargement of the affected sinuses performed in the operating room under general anesthesia.
  Arms: Endoscopic Sinus Surgery (ESS)
Other: General Anesthesia — ESS will be performed under general anesthesia in the operating room
  Arms: Endoscopic Sinus Surgery (ESS)
Other: Local and topical anesthesia — EPIC will be performed under topical and local anesthesia in a clinic setting
  Arms: Endoscopic polypectomy in clinic (EPIC)

SUMMARY:
Chronic rhinosinusitis, also called chronic sinusitis, is a very common life-long disease affecting over 5% of the Canadian population. Its symptoms, including daily facial pain and headache, an inability to breath through the nose and complete smell loss, regularly impair one's ability to work and to enjoy and participate in daily activities. The annual cost of chronic sinusitis to Canada is estimated at $1.3 billion while the government pays an estimated $860 million yearly for chronic sinusitis treatment. Chronic sinusitis with polyps, the most common type of chronic sinusitis, is usually treated with a combination of medications and surgery. Until now, surgical treatment has only been performed in the operating room, at a cost of about $3500 per procedure. But, recent studies have shown that a new procedure, "in-clinic polyp removal", can provide an improvement in patient symptoms to levels equal to those for sinus surgery performed in a hospital operating room. Moreover, in clinic polyp removal has additional advantages including a shorter procedure recovery time, a significantly lower cost to the health care system (about one-tenth the cost or $450), and a shorter wait time for treatment. With the proposed pragmatic trial, the investigators will determine whether the in clinic polyp removal procedure is as good as sinus surgery in the operating room at controlling patient symptoms of chronic sinusitis. The investigators will also determine the cost and health-benefits for a patient, the healthcare system and for society of in clinic polyp removal in comparison to sinus surgery done in a hospital operating room. The investigators will then know if this new treatment, in clinic polyp removal, can replace sinus surgery as the standard of care for these patients.

DETAILED DESCRIPTION:
Chronic rhinosinusitis (CRS) is common, with a Canadian prevalence of 5%, and associated with significant morbidity having a health state utility value equivalent to end-stage renal disease. Understandably, CRS impairs workplace productivity but that productivity substantially increases following surgical treatment.

However, the wait time to receive surgical treatment (ESS) maybe up to 8 months or longer, with a cost to the Government of $3500/ESS procedure. The annual direct cost of CRS is estimated at $860 million with an overall financial impact of 1.3 billion dollars per year for Canada. Endoscopic polypectomy in clinic (EPIC), a potential disruptive innovation, is a drastically deescalated form of ESS performed in clinic instead of the operating room. EPIC appears to provide quality of life (QofL) improvement equivalent to that reported for ESS. EPIC has a shorter wait time and lower cost to a government, i.e. nearly one-tenth of ESS or about $450. A pilot economic evaluation study demonstrated that EPIC was cost-effective compared to ESS. This has created a controversy about which treatment should be employed for these patients. Further, a recent Cochrane review identified the need for high-quality randomised controlled trials to determine if ESS has additional benefit over polypectomy as there is currently insufficient evidence to draw conclusions about the superiority of polypectomy or ESS for the management of CRS with polyps.

The proposed national multicenter randomised controlled trial will determine whether EPIC is non-inferior to the current treatment standard, ESS, in QofL improvement for patients with CRS with polyps. It will also assess the cost-effectiveness of performing EPIC in place of ESS. The investigators hypothesize that EPIC will be non-inferior to ESS for QofL improvement while reducing health care cost. This would imply that EPIC is a dominant strategy and that the ESS strategy represents over-treatment in this patient population. The study findings would position EPIC into the current CRS treatment paradigm thereby transforming care and reducing costs both nationally and internationally.

ELIGIBILITY:
Inclusion Criteria:

1. Age 18 years or older
2. Diagnosis of chronic rhinosinusitis with polyps requiring surgical treatment after having been treated with medical therapy as designated by the Canadian clinical practice guidelines for acute and chronic sinusitis. 15
3. Bilateral nasal polyps present of Grade ≥ 2 on each side as determined by the Lildholdt scale score measured by nasal endoscopy at the screening visit.
4. Must have nasal blockage score greater than or equal to 2 on the sinonasal outcome test SNOT-22 at the screening visit.
5. Must have an American Society of Anesthesiologists physical status PS3 classification or less.
6. Participants with comorbid asthma or chronic obstructive pulmonary disease (COPD) must have stable disease with no exacerbations (no emergency room visits, hospitalisations, or oral or parental steroid use for these lower respiratory conditions) within 3 months before the screening visit.
7. Must be capable, in the opinion of the investigator, of providing informed consent to participate in the study. Participants must sign an informed consent document indicating that they understand the purpose of and procedures of the study and are willing to participate in the study.

Exclusion Criteria:

1. Women who are pregnant or breast feeding as per patient's report
2. Patients with hyperplastic polyps or polyps large enough that they result in external nasal deformity
3. Facial pain/pressure score higher than 2 on the sinonasal outcome test SNOT-22 at the screening visit.
4. History of any surgical procedure that prevents the ability to accurately grade the nasal polyps
5. Participants who will not be able to complete the follow-up appointments/evaluations
6. Have significant oral structural abnormalities, e.g. unrepaired cleft palate
7. Septal deviation requiring correction in order to perform either EPIC or ESS procedures
8. Diagnosis of an immunodeficiency or immunocompromised state
9. Diagnosis of cystic fibrosis
10. Diagnosis of allergic fungal sinusitis
11. Contraindication to the use of oral corticosteroids (e.g. uncontrolled diabetes, congestive heart failure, uncontrolled hypertension, known renal insufficiency, known peptic ulcer disease, known glaucoma, pregnancy)
12. History of either Churg-Strauss syndrome, primary ciliary dyskinesia, or vasculitis (e.g. granulomatosis with polyangiitis(GPA))
13. Allergy, hypersensitivity, or contraindication to the use of local or topical lidocaine anesthetics, nasal topical 1:1000 adrenaline, nasal decongestants, nasal steroid spray
14. Any serious or unstable concurrent disease, psychiatric disorder, or any significant condition that, in the opinion of the investigator, could confound the results of the study or could interfere with the participant's participation or compliance with the study
15. A recent (within 1 year of the screening visit) clinically significant history of drug or alcohol abuse, or dependence that, in the opinion of the investigator could interfere with the participant's participation or compliance with the study
16. Inability to read and understand English
17. Any medical condition that in the opinion of the investigator would interfere with the treatment
18. Any participant who is unfit to undergo surgery under general anesthesia
19. Current participation in another clinical trial at the time of the screening visit.
20. Participant is unable to undergo an awake procedure
21. Diagnosis or Aspirin Exacerbated Respiratory Disease (AERD)

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 140 (Estimated)
Dates: Start 2017-04-11 (Actual); Primary Completion 2025-12 (Estimated); Study Completion 2026-12 (Estimated)

PRIMARY OUTCOMES:
Sinonasal Outcome Test-22 (SNOT-22) | 3 months

SECONDARY OUTCOMES:
Peak Nasal Inspiratory Flow (PNIF): | 3 months
Iowa Satisfaction with Anesthesia Scale (ISAS) | 3 months
  Patient satisfaction with anesthesia for the treatment procedure
Work Productivity and Activity Impairment: Specific Health Problem (WPAI:SHP) | 3 months
  Work Impairment related to chronic rhinosinusitis
EQ-5D-5L | 3 months
  Quality of Life
Participant Health Resource Consumption Survey | 3 months
  Individual Health Resource Consumption
Adverse Events | 3 months

OTHER OUTCOMES:
Lund-Kennedy Endoscopic Scoring Scale | 3 months
  Endoscopic inflammation of the nose and paranasal sinuses after treatment
Visual Analogue Scale (VAS) for satisfaction with assigned procedure | 3 months
  Satisfaction with assigned procedure

CONTACTS AND LOCATIONS:
Overall Officials: Shaun Kilty, MD, Principal Investigator — The Ottawa Hospital Research Institute
Locations (4):
- Canada (4):
  - Vancouver General Hospital, Vancouver, British Columbia
  - St. Joseph's Hospital London, London, Ontario
  - Ottawa Hospital Research Institute, Ottawa, Ontario
  - McGill University Health Center, Montreal, Quebec

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Kilty S, Thavorn K, Janjua A, Lee J, MacDonald K, Meen E, Micomonaco D, Rotenberg B, Sowerby LJ, Tewfik M, Adams S, Frenette H, Lasso A, Fergusson DA. Endoscopic polypectomy performed in clinic for chronic rhinosinusitis with nasal polyps: study protocol for the EPIC multicentre randomised controlled trial. BMJ Open. 2020 Dec 2;10(12):e042413. doi: 10.1136/bmjopen-2020-042413. PMID 33268434